CLINICAL TRIAL: NCT03371134
Title: Role of Hypoxia Inducible Factor-1α (HIF-1α) in Skeletal Muscle Aging
Brief Title: Role of HIF-1α in Skeletal Muscle Aging
Acronym: HIF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: HIF
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Satellite cells isolated from muscular biopses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcopenic group: Harvesting of muscular biopsies Muscular biopsies will be harvested from old sarcopenic patients undergoing hip replacement surgery
  Interventions: Biological: Harvesting of muscular biopsies
- Control group: Harvesting of muscular biopsies Muscular biopsies will be harvested from young patients undergoing Anterior Cruciate Ligament (ACL) reconstruction surgery
  Interventions: Biological: Harvesting of muscular biopsies

INTERVENTIONS:
Biological: Harvesting of muscular biopsies — Muscular biopsies will be harvested during surgery; them satellite cells will be isolated and characterized in vitro.

SUMMARY:
Deficits in skeletal muscle function exist during aging and muscular dystrophy, and suboptimal function has been related to factors such as atrophy, excessive inflammation and fibrosis. Sarcopenia is the age-related loss of skeletal muscle mass and function. It is now recognised as a major clinical problem for older people and research in the area is expanding exponentially. This interest stems from the fact that sarcopenia is both common and associated with serious health consequences in terms of frailty, disability, morbidity and mortality. The age-related loss of human skeletal muscle mass is due to a decrease in myofibre size and number with the loss of both fast and slow type myofibres, although the loss of fast myofibres tends to start earlier, at ∼70 years. Many factors influence the decrease in muscle mass. A significant contributor is an anabolic resistance of older skeletal muscle to protein nutrition as seen during immobilisation which can be ameliorated at least in part by resistance exercise and dietary supplementation. Other intensive areas of research are related to the loss of innervation and oxidative damage. Moreover, ineffective muscle regeneration underlies each condition and has been attributed to a deficit in myogenic potential of resident stem cells or satellite cells. It is now widely accepted that satellite cells, and generally adult stem cells, are normally quiescent and tend to reside in hypoxic areas of the tissue to preserve their undifferentiated state. To govern these processes, cells have developed a very complex machinery that is mainly regulated by a group of transcription factors known as hypoxia-inducible factors (HIFs). In particular, several observations support the idea that oxygen deprivation and HIF-1a may play a key role during ischemia to activate the regeneration process, which, after an initial hypoxic insult, needs to proceed under normoxia. On these bases, in this study we will investigate the role of HIF-1a in skeletal atrophy during aging.

DETAILED DESCRIPTION:
Deficits in skeletal muscle function exist during aging and muscular dystrophy, and suboptimal function has been related to factors such as atrophy, excessive inflammation and fibrosis. Sarcopenia is the age-related loss of skeletal muscle mass and function. It is now recognised as a major clinical problem for older people and research in the area is expanding exponentially. This interest stems from the fact that sarcopenia is both common and associated with serious health consequences in terms of frailty, disability, morbidity and mortality. The age-related loss of human skeletal muscle mass is due to a decrease in myofibre size and number with the loss of both fast and slow type myofibres, although the loss of fast myofibres tends to start earlier, at ∼70 years. Many factors influence the decrease in muscle mass. A significant contributor is an anabolic resistance of older skeletal muscle to protein nutrition as seen during immobilisation which can be ameliorated at least in part by resistance exercise and dietary supplementation. Other intensive areas of research are related to the loss of innervation and oxidative damage. Moreover, ineffective muscle regeneration underlies each condition and has been attributed to a deficit in myogenic potential of resident stem cells or satellite cells. It is now widely accepted that satellite cells, and generally adult stem cells, are normally quiescent and tend to reside in hypoxic areas of the tissue to preserve their undifferentiated state. To govern these processes, cells have developed a very complex machinery that is mainly regulated by a group of transcription factors known as hypoxia-inducible factors (HIFs). In particular, several observations support the idea that oxygen deprivation and HIF-1a may play a key role during ischemia to activate the regeneration process, which, after an initial hypoxic insult, needs to proceed under normoxia. On these bases, in this study we will investigate the role of HIF-1a in skeletal atrophy during aging.

In particular, we will isolate satellite cells from muscular biopsies harvested from old sarcopenic patients and from young patients. The, we will measure HIF-1a levels and we will compare them.

ELIGIBILITY:
Inclusion Criteria:

* Sarcopenic patients (measured by DXA) affected by hip osteoarthritis, developmental dysplasia of the hip or hip fracture and undergoing hip replacement surgery (for the sarcopenic group)
* Patients affected by traumatic ACL tears and undergoing ACL reconstruction surgery (for the control group)
* Patients between 18 and 35 years old (for the control group)
* Patients between 65 and 90 years old (for the sarcopenic group)
* 18 ≤ Body Mass Index (BMI) ≤ 30 kg/m2

Exclusion Criteria:

* Diseases that can affect bone or muscle metabolism
* Pharmacological therapies that can interact with bone or muscle metabolism
* Bone metastases
* Bone infections
* HIV, hepatitis B virus, hepatitis C virus or Treponema pallidum positivity
* BMI ≥30kg/m2

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be selected and evaluated in the primary care clinic. The eligibility criteria will be checked 2-4 weeks before surgery.
  Muscular biopsies will be harvested from discarded material during surgery.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2018-01-10 (Estimated); Primary Completion 2019-01-10 (Estimated); Study Completion 2020-07-26 (Estimated)

PRIMARY OUTCOMES:
Evaluation of HIF-1a expression levels in satellite cells isolated from sarcopenic and young | 1 year
  Western blot analysis of HIF-1a levels and of its downstream targets (Vascular Endothelial Growth Factor: VEGF, phosphoglycerate kinase: PGK, Prolylhydroxilases: PHD2)

SECONDARY OUTCOMES:
Evaluation of sarcopenic profile in satellite cells harvested from old sarcopenic patients | 6 months
  Real Time polymerase chain reaction: PCR analysis of MURF1 and atrogin1 (markers of muscular aging)
Correlation of HIF-1a levels with the degree of sarcopenia in the satellite cells of old sarcopenic patients | 1 year
  chromatin immunoprecipitation: ChiP seq analysis of HIF-1a downstream targets
Evaluation of differences in satellite cells number between young and old patients | 6 months
  To evaluate differences in cell number two different immunohistochemical analyses will be used in order to obtain a ratio: 1. Immunofluorescence for PAX7 (satellite cell markers) and 2. BrdU will be performed and the ration between PAX7 positive cells and bromodeoxyuridine: BrdU positive cells will be calculated.
Evaluation of HIF-1a stabilization on satellite cells treated with PHDs inhibitors | 1 year
  Prolylhydroxilases: PHDs inhibitors (FG-4592 e PLG) will be tested in vitro to analyze HIF-1a downstream targets (Vascular Endothelial Growth Factor: VEGF, phosphoglycerate kinase: PGK, Prolylhydroxilases: PHD2) by real time PCR
Evaluation of satellite cell proliferation in cells treated with PHDs inhibitors | 1 year
  Prolylhydroxilases: PHDs inhibitors (FG-4592 e PLG) will be tested in vitro to analyze cell proliferation (RealTime Glow and CellTox kits)
Evaluation of satellite cell differentiation in cells treated with PHDs inhibitors | 1 year
  Prolylhydroxilases: PHDs inhibitors (FG-4592 e PLG) will be tested in vitro to analyze cell differentiation (Immunofluorescence and Realt Time PCR analysis for differentiation markers: MyoD, Myogenin and Myosin Heavy Chain)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mangiavini, Dr, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi

IPD SHARING:
Plan to Share IPD: No